CLINICAL TRIAL: NCT00387140
Title: A Randomized Double-blind, Placebo-and Active Comparator-Controlled 2-Part Study to Evaluate the Efficacy of MK2295 in Patients With Postoperative Dental Pain
Brief Title: A Study to Evaluate the Safety and Efficacy of an Investigational Drug in the Treatment of Postoperative Dental Pain (MK-2295-005)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2295-005; MK2295-005; 2006_518
Record Dates: First submitted 2006-10-09; First posted 2006-10-12 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Pain, Postoperative; Tooth Extraction
Keywords: Dental Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative; Toothache | interventions — MK-2295

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK2295

SUMMARY:
This study is being conducted to evaluate the safety and tolerability of the drug and to evaluate its efficacy compared to placebo and to ibuprofen in the treatment of postoperative dental pain in male patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients in generally good health who are scheduled to have two or more third molars removed, at least one of which is partially or completely embedded in bone and is a mandibular impaction

Exclusion Criteria:

* Patient has a temperature of 37.5C or greater prior to dosing
* Patient has participated in another clinical study within the last 4 weeks

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 89 (Actual)
Dates: Start 2006-10; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Peak analgesic response, safety, and tolerability | Over 24 Hours

SECONDARY OUTCOMES:
Onset of analgesia, duration of analgesia | Over 24 Hours

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC